CLINICAL TRIAL: NCT00732797
Title: Evaluation of the Cost-effectiveness of Booklet-based Self-management of Dizziness in Primary Care, With and Without Expert Telephone Support
Brief Title: A Trial of Booklet Based Self Management of Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PB-PG-0107-12069; 08/H0504/31
Record Dates: First submitted 2008-08-07; First posted 2008-08-12 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Dizziness
Keywords: Dizziness; Self-management; booklet-based; vestibular rehabilitation
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Care (No Intervention): Participants will receive routine care.
- Booklet (Active Comparator): Participants will receive self-treatment booklets, but no expert telephone support.
  Interventions: Behavioral: Self-treatment booklet
- Booklet &Therapist Support (Active Comparator): Participants will receive self-treatment booklets, and up to an hour's expert telephone support.
  Interventions: Behavioral: Self-treatment booklet; Behavioral: Remote telephone support

INTERVENTIONS:
Behavioral: Self-treatment booklet — A booklet outlining vestibular rehabilitation exercises
  Arms: Booklet; Booklet &Therapist Support
Behavioral: Remote telephone support — Up to an hour's remote support from an expert vestibular therapist
  Arms: Booklet &Therapist Support

SUMMARY:
The investigators primary aim is to test whether or not provision of the self-help booklet teaching VR exercises, with up to one hour of telephone support from a vestibular therapist, will be more effective than routine care in reducing symptoms in dizzy patients in primary care. The investigators will also explore the extent to which patients may benefit from the self-help booklet without support. The investigators will determine whether these models of delivery are less costly than routine care of dizzy patients, as they should reduce the number of patients seeking referral to secondary care for unnecessary assessments.

DETAILED DESCRIPTION:
Chronic dizziness has a prevalence of up to 25% in the community, and 1 in 10 working age adults and 1 in 5 older people report some degree of handicap due to dizziness. Dizziness can lead to reduced quality of life, anxiety and emotional distress, loss of fitness, unsteadiness and vulnerability to falling. Reviews of the management of dizziness have concluded that no medication has well-established value or is suitable for long-term use, and vestibular rehabilitation (VR) is now recommended as the treatment of choice. Professor Lucy Yardley has carried out trials showing that chronic dizziness can be treated effectively using a self-help booklet to teach patients vestibular rehabilitation exercises that promote neurological adaptation and skill and confidence in balance. These exercises are carried out for 10 minutes twice daily at home, and involve gently increasing the speed of making normal head movements. However, brief support from a trained nurse was provided in these trials, and this model of managing dizzy patients has not been taken up due to a lack of skills and resources in primary care.

We have received funding to evaluate the cost-effectiveness of two new models of delivery of vestibular rehabilitation. Our primary aim is to test the hypothesis that provision of the self-help booklet teaching vestibular rehabilitation exercises, with up to one hour of remote telephone support from an expert vestibular therapist, will be more effective than routine care in reducing symptoms (and therefore also disability and handicap) in dizzy patients in primary care. We will also explore the extent to which patients may benefit from provision of the self-help booklet without support. We will determine whether these models of delivery are less costly than routine care of dizzy patients, as they should reduce the number of patients seeking referral to secondary care for unnecessary assessments.

This trial involves patients taking part in either a 12 week self-treatment programme (with or without telephone support from an expert vestibular therapist) or routine care, and completing questionnaires before and after the self-treatment, and also one year later. We will recruit 330 participants with dizziness who are registered with 30 general practices around Southampton and Berkshire. The trial will be carried out approximately between June 2008 and June 2011.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or over
* Be registered with a participating GP
* Must have visited their GP for dizziness in the last 2 years
* Must complete the consent form, and baseline questionaire indicating they are still suffering from dizziness and that quick head movements make them dizzy.

Exclusion Criteria:

* Non-Labyrinthe cause of dizziness identified by GP
* Medical contraindications from making normal head movements
* Serious co-morbidity
* Moved away from practice
* Recently deceased
* Non-English speakers, and unable to read/write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Self-reported measures of dizziness | Measured at beseline, 12 weeks and 1 year.

SECONDARY OUTCOMES:
Quality of life effects of dizziness | Measured at baseline, 12 weeks and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Yardley, Principal Investigator — University of Sothampton
Locations (1):
- Hampshire PCT and Berkshire PCT, Southampton, United Kingdom

REFERENCES:
- [Derived] Muller I, Kirby S, Yardley L. Understanding patient experiences of self-managing chronic dizziness: a qualitative study of booklet-based vestibular rehabilitation, with or without remote support. BMJ Open. 2015 May 18;5(5):e007680. doi: 10.1136/bmjopen-2015-007680. PMID 25986639
- [Derived] Yardley L, Barker F, Muller I, Turner D, Kirby S, Mullee M, Morris A, Little P. Clinical and cost effectiveness of booklet based vestibular rehabilitation for chronic dizziness in primary care: single blind, parallel group, pragmatic, randomised controlled trial. BMJ. 2012 Jun 6;344:e2237. doi: 10.1136/bmj.e2237. PMID 22674920
- [Derived] Yardley L, Kirby S, Barker F, Little P, Raftery J, King D, Morris A, Mullee M. An evaluation of the cost-effectiveness of booklet-based self-management of dizziness in primary care, with and without expert telephone support. BMC Ear Nose Throat Disord. 2009 Dec 29;9:13. doi: 10.1186/1472-6815-9-13. PMID 20098640